CLINICAL TRIAL: NCT00102232
Title: Effect of Choline Supplemented as Phosphatidylcholine on Post-Methionine Loading and Fasting Concentrations of Plasma Homocysteine in Healthy Volunteers
Brief Title: Effect of Phosphatidylcholine on Plasma Homocysteine in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen Centre for Food Sciences (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: TNO4963
Record Dates: First submitted 2005-01-25; First posted 2005-01-26 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-01

CONDITIONS: Healthy; Cardiovascular Diseases
Keywords: phosphatidylcholine; choline; homocysteine; cardiovascular disease prevention; human; cardiovascular health
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Dietary Supplements; Phosphatidylcholines

INTERVENTIONS:
Procedure: supplementation with phosphatidylcholine

SUMMARY:
The purpose of this study is to determine whether supplementation with phosphatidylcholine lowers plasma homocysteine concentrations in healthy men.

DETAILED DESCRIPTION:
A high homocysteine concentration is a potential risk for cardiovascular disease. Plasma homocysteine concentrations can be lowered through betaine supplementation. However, effects of choline supplementation, the precursor for betaine, on plasma homocysteine concentrations in healthy humans are unknown. If supplementation with choline or phosphatidylcholine, the form in which choline occurs in foods, lowers homocysteine concentrations, then extra intake of these compounds may lower cardiovascular disease risk in humans.

Comparison: We compared the effects of supplementation with phosphatidylcholine to the effects of a placebo on fasting and post-methionine concentrations of plasma homocysteine in healthy men.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males as assessed by the health and lifestyle questionnaire, physical examination and results of the pre-study laboratory tests
* Body Mass Index (BMI) ≤ 33 kg/m2
* Normal Dutch eating habits, including use of breakfast
* Willing not to use supplements containing B-vitamins, lecithin, choline (derivatives) or betaine from the oral information session until the end of the study
* Voluntary participation
* Having given their written informed consent
* Willing to comply with the study procedures, including dietary restrictions
* Willing to accept use of all nameless data, including publication, and the confidential use and storage of all data
* Willing to accept the disclosure of the financial benefit of participation in the study to the authorities concerned

Exclusion Criteria:

* Participation in any clinical trial including blood sampling and/or administration of products up to 90 days before Day 01 of this study
* Participation in any non-invasive clinical trial up to 30 days before Day 01 of this study
* Having a history of medical or surgical events that may significantly affect the study outcome, including cardiovascular disease or hypertension
* Use of medication known to interfere with homocysteine metabolism
* Plasma total homocysteine concentrations > 26 µmol/L
* Plasma vitamin B6 concentrations ≤ 15 nmol/L
* Serum vitamin B12 concentrations < 138 pmol/L
* Serum folic acid concentrations < 5.0 nmol/L
* Alcohol consumption > 28 units/week
* Reported unexplained weight loss or gain of > 2 kg in the month prior to the pre-study screening
* Reported slimming or medically prescribed diet
* Reported food allergy
* Reported vegan or macrobiotic
* Use of B-vitamin supplements, lecithin, or supplements containing choline (derivatives) or betaine, more than once weekly < 1 month before screening
* Recent blood or plasma donation (< 1 month prior to the start of the study)
* Not willing to stop blood or plasma donation during the study
* Personnel of TNO Nutrition and Food Research, their partner and their relatives in the first and second remove
* Not having a general practitioner
* Not willing to accept information-transfer concerning participation in the study, or information regarding his/her health, like laboratory results, findings at anamnesis or physical examination and eventual adverse events to and from his general practitioner

Ages: 50 Years to 71 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26
Dates: Start 2003-05; Study Completion 2003-07

PRIMARY OUTCOMES:
Concentrations of plasma homocysteine in the fasting state
Concentrations of plasma homocysteine after a methionine load

SECONDARY OUTCOMES:
Lipid concentrations
Liver enzymes
Creatinine
B-vitamins

CONTACTS AND LOCATIONS:
Overall Officials: Petra Verhoef, PhD, Study Chair — Wageningen Centre for Food Sciences; Elizabeth J Brink, PhD, Principal Investigator — TNO Nutrition and Food Research
Locations (2):
- Netherlands (2):
  - Wageningen Centre for Food Sciences, Wageningen
  - TNO Nutrition and Food Research, Zeist